CLINICAL TRIAL: NCT03960268
Title: A Pilot Study of Safety and Biomarkers In Hidradenitis Suppurativa Participants Receiving Brodalumab
Brief Title: Biomarkers In Hidradenitis Suppurativa Participants Receiving Brodalumab
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Valeant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JFR-0989
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Acne Inversa; Brodalumab
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — brodalumab

STUDY DESIGN:
Intervention Model Description: Open Label Single Arm Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Brodalumab 210mg subcutaneously every 2 weeks for 24 weeks
  Interventions: Drug: Brodalumab

INTERVENTIONS:
Drug: Brodalumab — interleukin 17 receptor A antagonist
  Other Names: Siliq

SUMMARY:
Phase 0 Study of Brodalumab in patients with moderate to severe Hidradenitis Suppurativa to identify biomarkers of disease activity and clinical response.

DETAILED DESCRIPTION:
Phase 0, Open Label study of Brodalumab in patients with moderate to severe Hidradenitis Suppurativa. Consisting of n=10 patients receiving 210mg subcutaneously every 2 weeks for 24 weeks. Patients will be followed for a period of 36 weeks (12 weeks after last dose of Brodalumab) to assess for safety.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diagnosis of Hidradenitis Suppurativa by the PI
* Age 18 or older
* Moderate to Severe Hidradenitis Suppurativa as determined by the PI

Exclusion Criteria:

* Inflammatory Bowel Disease
* HIV Positive
* Active Hepatitis B or C Infection
* Pregnant or Breastfeeding
* no concurrent use of any systemic antibiotics/retinoids/imunosuppressants (require washout period of >5 half lives)
* Any medical, psychological or social condition that, in the opinion of the investigator, would jeopardize the health or well being go the participant during any study procedures or the integrity of the data
* High Suicide Risk as determined by the Columbia Suicide Severity Rating Scale
* History of Keloid Scarring

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Biomarkers at Week 12 | Week 12 compared with baseline.
  Primary Outcomes would be the change in lesional tissue levels of IL-17A, IL-17C, IL-17F and IL-23 measured in pg/mL measured in pg/mL
Biomarkers at Week 24 | Week 24 compared with baseline.
  Primary Outcomes would be the change in lesional tissue levels of IL-17A, IL-17C, IL-17F and IL-23 measured in pg/mL measured in pg/mL
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Week 0 to Week 24
  Incidence of Grade 2/3 adverse events during the study

SECONDARY OUTCOMES:
Clinical Response at Week 12 (as measured by HiSCR) | Week 12 compared with Baseline
  Clinical Response compared to baseline as assessed by the HiSCR (Hidradenitis Suppurativa Clinical Response) Defined as a greater than or equal to 50% reduction in inflammatory lesion count (abscesses plus inflammatory nodules), and no increase in abscesses or draining fistulas at Week 12 when compared with baseline
Clinical Response at Week 12 (as measured by modified Sartorius Score) | Week 12 compared with Baseline
  Clinical Response compared to baseline as assessed by the modified Sartorius Score as follows: Sum of separate scoring for each affected area using the data recorded as follows: a) 3 points per anatomical region involved; b) 6 points for each fistula and 1 point for each nodule or abscess; c) 1 point when the longest distance between two relevant lesions in each affected area is <5 cm; 3 points when it is 5-10 cm; and 9 points when it is >10 cm; d) 9 points when there is no clear separation of lesions from adjacent normal skin and 0 points when there is.
Clinical Response at Week 12 (as measured by IHS4) | Week 12 compared with Baseline
  Clinical Response compared to baseline as assessed by IHS4 (International Hidradenitis Suppurativa Severity Score) using the scoring system as follows: Total= (Number of nodules x1) + (Number of abscesses x2) + (Number of draining sinuses/fistulae x4)
Clinical Response at Week 24 (as measured by HiSCR) | Week 24 compared with Baseline
  Clinical Response compared to baseline as assessed by the HiSCR (Hidradenitis Suppurativa Clinical Response) Defined as a greater than or equal to 50% reduction in inflammatory lesion count (abscesses plus inflammatory nodules), and no increase in abscesses or draining fistulas at Week 24 when compared with baseline
Clinical Response at Week 24 (as measured by modified Sartorius Score) | Week 24 compared with Baseline
  Clinical Response compared to baseline as assessed by the modified Sartorius Score as follows: Sum of separate scoring for each affected area using the data recorded as follows: a) 3 points per anatomical region involved; b) 6 points for each fistula and 1 point for each nodule or abscess; c) 1 point when the longest distance between two relevant lesions in each affected area is <5 cm; 3 points when it is 5-10 cm; and 9 points when it is >10 cm; d) 9 points when there is no clear separation of lesions from adjacent normal skin and 0 points when there is.
Clinical Response at Week 24 (as measured by IHS4) | Week 24 compared with Baseline
  Clinical Response compared to baseline as assessed by IHS4 (International Hidradenitis Suppurativa Severity Score) using the scoring system as follows: Total= (Number of nodules x1) + (Number of abscesses x2) + (Number of draining sinuses/fistulae x4)

CONTACTS AND LOCATIONS:
Overall Officials: John W Frew, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller Unviersity, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navrazhina K, Frew JW, Gilleaudeau P, Sullivan-Whalen M, Garcet S, Krueger JG. Epithelialized tunnels are a source of inflammation in hidradenitis suppurativa. J Allergy Clin Immunol. 2021 Jun;147(6):2213-2224. doi: 10.1016/j.jaci.2020.12.651. Epub 2021 Feb 3. PMID 33548397